CLINICAL TRIAL: NCT01685385
Title: B-type NAtriuretic Peptide In Critically Ill : A Multicentric Diagnostic Study (B-rAPID)
Acronym: B-RAPID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahatma Gandhi Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Rajnish joshi, Dr.Rajnish Joshi, Mahatma Gandhi Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MGIMS001/2012
Record Dates: First submitted 2012-09-08; First posted 2012-09-14 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Heart Failure; Congestive Cardiac Failure; Dyspnoea
Keywords: Dyspnoea; BNP; Chronic heart failure; congestive heart failure
MeSH Terms: conditions — Heart Failure; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diagnostic intervention group A (Active Comparator): Patients who will receive the BNP test
  Interventions: Other: Patients who will receive the BNP test
- Group B (No Intervention): Patients who will not receive the BNP test.

INTERVENTIONS:
Other: Patients who will receive the BNP test — Patients in Diagnostic Intervention Group A will receive the point-of-care BNP test, in addition to all other diagnostics they receive in addition
  Arms: Diagnostic intervention group A

SUMMARY:
Difficulty in breathing or increased rate of breathing are common causes of admission to intensive care unit. This may be due to heart failure, or other causes such as infection in the lungs. Treating doctors usually perform Chest X-ray, ECG, and other tests to know if breathlessness is due to heart failure or other cause. Doctors also give medicines to treat heart failure, or other conditions of the lungs based on the symptoms and investigation results. BNP is released by heart which is not functioning well. However BNP levels are also high in case of severe infection.Hence there is equipoise in utility of BNP measurements among critically ill patients, and it is not a current standard of care. The current cost of this test (about 1000 rupees per measurement) is high, and hence its utility needs to be carefully examined before a widespread use. The investigators intend to test the hypothesize that that on-admission BNP measurements, help clinicians identify CHF early, which may modify therapeutic decisions, and improve outcomes. The current study is designed with an objective to determine if on-admission BNP value and availability of its test results to treating physicians will reduce in-hospital, and 30-day mortality and in-hospital morbidity.

DETAILED DESCRIPTION:
There usually remains a diagnostic uncertainty as differentiation between cardiogenic or non-cardiogenic cause of dyspnea. Often there are multiple underlying etiologies for acute onset dyspnea, and their evaluation leads to diagnostic delays, and hence longer hospital stay. While various clinical symptoms, signs and imaging based investigations are used in this differentiation, their accuracy remains low, and overlapping features preclude such differentiation. Echocardiography is an important adjunct in making such differentiation, but operator skill, and lack of availability of this technique at point of care are barriers in use of this modality. B-type natriuretic peptide (BNP), a rapidly-assayed, serum biomarker, has been found to be effective in distinguishing congestive heart failure (CHF) from other causes of dyspnea in the emergency or urgent care settings. Recently this test has become available at point of care (Alere Heart-Check). Ease, low cost, and objectivity in measurement of BNP has led to widespread incorporation of BNP and its precursor NT-pro-BNP into the clinical evaluation of CHF.

Circulating levels of BNP/NT-proBNP are normally very low in healthy individuals. In response to increased myocardial wall stress due to volume- or pressure-overload states (such as in CHF), the BNP gene is activated in cardiomyocytes. This results in the production of an intracellular precursor propeptide (proBNP108); further processing of this propeptide results in release of the biologically inert aminoterminal fragment (NT-proBNP) and the biologically active BNP.Various studies have been performed to determine cut-off level to make a differentiation between presence or absence of CHF using this test. BNP level below 50pg/ml rules out CHF with a negative predictive value of 96%. (3) In the same study by Maisel et al the diagnostic accuracy of B-type natriuretic peptide to rule in CHF at a cutoff of 100 pg per milliliter or more was 83.4 percent. However subsequent studies have instead suggested a multiple cut-point strategy (Less than 100pg/ml rules out CHF (NPV 90%), more than 400 pg/ml rules in CHF (91% specificity) while intermediate values representing a grey zone. Individuals with renal dysfunction have elevated BNP levels, and a lower cut-off to exclude CHF in such patients is 200pg/ml. Individuals with a high BMI have falsely low levels and a BMI adjusted correction is used (Lower cut-off of 54pg/mL if BMI >35kg/m2). The levels of BNP as well as NT-Pro-BNP have similar elevations in CHF, later being three times as much higher. (1) Use of BNP to differentiate CHF from other causes of dyspnea, (4) and ease in its measurement has resulted in increase in its use in intensive care settings, as point-of-care testing has a potential to change outcomes. However when the test is used in this setting, very high BNP levels were detected in critically ill patients with sepsis and shock. In patients with shock, levels below 1200pg/ml had a negative predictive value of 92% for cardiogenic shock. Such high levels in patients with compromised systolic function have questioned utility of this measure to distinguish between CHF and other causes in critical care settings. It is debated that in critically ill patients, coexisting other organ dysfunction, rapid changes in volume status, variable bioavailability and burst synthesis of BNP may all confound interpretation of BNP levels. However despite this confounding, even in critically ill patients higher values are associated with adverse prognosis, and very low levels (less than 100pg/ml) will mean a preserved left ventricular function. Thus, while it is known that BNP really gives useful information, not already available from other clinical, radiologic and biochemical measurements, what the investigators do not know is if the test results become available in an intensive care unit setting, will it help treating physicians to make meaningful clinical decisions.

Given above considerations, there is equipoise in utility of BNP measurements among critically ill patients, and it is not a current standard of care. The current cost of this test (about 1000 rupees per measurement) is high, and hence its utility needs to be carefully examined before a widespread use. The investigators intend to test the hypothesize that that on-admission BNP measurements, help clinicians identify CHF early, which may modify therapeutic decisions, and improve outcomes. The current study is designed with an objective to determine if on-admission BNP value and availability of its test results to treating physicians will reduce in-hospital, and 30-day mortality and in-hospital morbidity.

ELIGIBILITY:
Inclusion Criteria:

We will include all consecutive patients admitted to intensive care units in participating sites with all of the following features:

* Adult aged 18 years or more
* Acute onset dyspnea (duration 3 days or less) , defined as respiratory rate of 20 or more.
* Treating physician considers patient to be critically ill so as to warrant care in intensive care unit.

Exclusion Criteria:

Patients for whom consent is not obtained will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | From admission to death in hospital and upto 30 days after admission to the hospital, whichever is earlier
  Assessment of In hospital mortality within 30-days of admission, and comparison between groups A and B.
30-day mortality | Upto 30 days from admission to hospital
  Mortality will be assessed after discharge from the hospital and upto 30 days from hospital admission and compared between groups A and B

SECONDARY OUTCOMES:
In-hospital morbidity | Time of admission to ICU till death or discharge or 30days after admission, whichever is earlier
  In-hospital morbidity, measured as a) duration of ICU stay, duration of hospital stay, need for mechanical ventilation or renal replacement during hospitalization, measured upto 30-days after admission to hospital

OTHER OUTCOMES:
Intensity of In-hospital therapies administered | First 24 hrs of ICU stay
  To compare the difference in cumulative dose of diuretics, parenteral antibiotics, corticosteroids, and bronchodilators administered within first 24 hours of admission to ICU, between groups A and B.
Time to initiate heart failure specific therapies | During hospital stay and upto 30-days after admission to hospital
  To Compare the difference in time to initiate heart failure specific therapies (diuretics, angiotensin converting enzyme inhibitors, beta-blockers, and spironolactone) in groups A and B, during hospital stay and upto 30-days of admission to hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Rajnish Joshi, MD, Principal Investigator — Sikkim Manipal Institute of Medical Sciences; Dr.Vishakha Jain, MD, Principal Investigator — Mahatma Gandhi Institute of Medical Science
Locations (4):
- India (4):
  - Assam Medical College, Dibrugarh, Assam
  - Jawaharlal Nehru Medical college, Wardha, Maharashtra
  - Mahatma Gandhi Institute of Medical Sciences, Wardha, Maharashtra
  - Sikkim Manipal Institute of Medical Sciences, Gangtok, Sikkim